CLINICAL TRIAL: NCT03372629
Title: A Two-part Single-center, Phase 1 Study to Assess the Tolerability, Safety, Pharmacokinetics (Including Food Interaction), and Pharmacodynamics of Ascending Single and Multiple Doses of ID-085 in Healthy Subjects
Brief Title: A Study to Evaluate if ID-085 is Safe, Its Fate in the Body as Well as Its Potential Effects on the Body in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-085-101; 2017-004124-30 (EudraCT Number)
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ID-085, single ascending dose (Part A) (Experimental): ID-085 administered at different single dose levels in a sequential manner, and in a maximum of 6 dose levels starting from 10 mg (number of cohorts and dose levels will depend on the safety and pharmacokinetic results of the previous cohort)
  Interventions: Drug: ID-085
- Placebo, single ascending dose (Part A) (Placebo Comparator): Matched placebo administered as single ascending doses in parallel to ID-085
  Interventions: Drug: Placebo oral capsule
- ID-085 multiple ascending dose (Part B) (Experimental): ID-085 administered in a twice daily (b.i.d.) dosing regimen at multiple dose levels. The starting dose will be either 10 or 30 mg and will be selected on the basis of the safety and pharmacokinetic results of the part A
  Interventions: Drug: ID-085
- Placebo, multiple ascending dose (Part B) (Placebo Comparator): Matched placebo administered as single ascending doses in parallel to ID-085
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ID-085 — Hard gelatin capsules for oral administration formulated in strengths of 10 mg, 100 mg, and 200 mg
  Arms: ID-085 multiple ascending dose (Part B); ID-085, single ascending dose (Part A)
Drug: Placebo oral capsule — Placebo capsules matching ID-085 capsules
  Arms: Placebo, multiple ascending dose (Part B); Placebo, single ascending dose (Part A)

SUMMARY:
The objective of this study is to evaluate the tolerability, safety, and pharmacokinetic of single- and multiple-ascending doses of ID-085 in healthy subjects.

DETAILED DESCRIPTION:
The study is designed in two parts, A and B.

Part A: single-center, double-blind, randomized, placebo-controlled, single ascending dose.

Part B: single-center, double-blind, randomized, placebo-controlled, multiple ascending dose.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Healthy male subjects for Part A, healthy male and female subjects for Part B aged between 18 and 55 years (inclusive) at screening.
* No clinically significant findings on physical examination at screening.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at screening.

Exclusion Criteria:

* History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Pregnant or lactating women.
* Known allergic reactions or hypersensitivity to the study treatment or drugs of the same class, or any of the excipients.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in PQ/PR interval (ms) | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  ECG variables are to be recorded using a standard 12-lead ECG
Changes from baseline in QRS interval (ms) | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  ECG variables are to be recorded using a standard 12-lead ECG
Changes from baseline in QT corrected for Bazett's formula (QTcB) interval (ms) | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  ECG variables are to be recorded using a standard 12-lead ECG
Changes from baseline in RR interval (ms) | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  ECG variables are to be recorded using a standard 12-lead ECG
Changes from baseline in heart rate (bpm) | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  ECG variables are to be recorded using a standard 12-lead ECG
Changes from baseline in supine systolic blood pressure | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  mm Hg
Changes from baseline in supine diastolic blood pressure | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  mm Hg
Changes from baseline in supine pulse rate | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  bpm
Changes from baseline in body weight | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  kg
Number of patients with treatment-emergent AEs and SAEs for each treatment period | up to 48 hours post-dose (Part A); up to Day 10 (Part B)
  Treatment-emergent AEs and treatment-emergent serious AEs

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to Day 3 (Part A), up to Day 10 (Part B)
Time to reach Cmax (tmax) | up to Day 3 (Part A), up to Day 10 (Part B)
Terminal half-life [t(1/2)] | up to Day 3 (Part A), up to Day 10 (Part B)
Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) | up to Day 3 (Part A), up to Day 10 (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Covance Clinical Research Unit - Clinical Pharmacology Services, Leeds, United Kingdom